CLINICAL TRIAL: NCT00537667
Title: A Single Centre, Open-Label, Randomised, Study to Evaluate the Effect of Anakinra (r-metHuIL-1ra) Alone and in Combination With PEGylated Recombinant Methionyl Human Soluble Tumour Necrosis Factor Receptor Type I (PEG sTNF-RI) on Synovial Inflammation in Subjects With Rheumatoid Arthritis.
Brief Title: The SPECTRA Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The safety profile of combination therapy became unacceptable.
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Organization: Swedish Orphan Biovitrum (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20000211
Record Dates: First submitted 2007-09-27; First posted 2007-10-01 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
Keywords: IL-1ra; PEG sTNF-RI; Synovial biopsy; Inflammation; Bone and Cartilage Destruction; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

ARMS (2):
- A (Active Comparator): anakinra
  Interventions: Drug: anakinra
- B (Experimental): anakinra and PEGsTNF-R1
  Interventions: Drug: anakinra and PEG sTNF-R1

INTERVENTIONS:
Drug: anakinra — anakinra
  Arms: A
Drug: anakinra and PEG sTNF-R1 — anakinra and PEG sTNF-R1
  Arms: B

SUMMARY:
The purpose of this study is to compare IL-1ra and the combination of IL-1ra and PEGsTNF-RI with respect to their ability to reduce inflammation and bone and cartilage destruction in the synovium of subjects with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA as determined by American College of Rheumatology (ACR) criteria (Appendix C)
* Disease duration of no less than 12 weeks of diagnosis confirmed by physician and source documentation
* Disease duration < 10 years
* Active RA at baseline as defined by a minimum of 6 or more swollen joints and 9 or more tender/painful joints (based on a 66/68-joint count excluding distal interphalangeal joints) at screening and baseline,

And

* C-reactive protein (CRP) > 2 mg/dL at screening.
* Have active clinical synovitis in the knee as determined by the investigator based on clinical evaluation
* 18 years of age or older
* Men or non-pregnant (negative serum HCG at screening unless surgically sterile or postmenopausal), non-breast-feeding women may be enrolled. Females of childbearing potential and males must use adequate contraceptive precautions as determined by the principal investigator.
* Subjects that have taken any DMARD for less than 3 months must not have taken DMARDs within 4 weeks prior to screening. Subjects that have taken any DMARD for longer than 3 months must not have taken DMARDs within 6 months of screening.
* Subject's doses of NSAIDs and oral corticosteroids (10 mg/day of prednisone or equivalent) must have been kept stable for 4 weeks before screening
* Subjects must not have had intrarticular injections in the joint that will be arthroscoped for at least 3 months prior to screening.

Before any study specific procedure or screening is done, the subject or legally acceptable representative must give informed consent for participation in the study (see Section 12.2). Before buccal smears and blood samples are taken for genetic testing, the subject or legally acceptable representative must give informed consent for use of those samples for genetic testing (see Section 12.2).

Exclusion Criteria:

* ACR functional class IV or American Rheumatology Association anatomical stage IV (see Appendix C)
* Disease duration >10 years
* Diagnosed with the following:

Felty's syndrome

Advanced or uncontrolled Diabetes Mellitus (defined as: HbA1c > 8%, peripheral neuropathy, renal/retinal involvement, or vascular disorders)

Malignancy, other than basal cell carcinoma of the skin or in situ carcinoma of the cervix, within the past five years

Any other major chronic inflammatory disease or syndrome (e.g., psoriatic arthritis, spondyloarthropathy, inflammatory bowel disease, fibromyalgia that required treatment in the last year)

* Any uncontrolled, clinically significant systemic disease
* Pre-existing or recent onset central nervous system demyelinating disorders
* Significant hematologic abnormalities
* A history of drug or alcohol abuse within the previous 24 weeks
* Known to be hepatitis B surface antigen, hepatitis C virus or Human Immunodeficiency Virus positive
* Any disorder that compromises ability to give informed consent for participation in this study
* Is expected to require a major surgical operation while on study that would interfere with the collection of the required assessments.
* Has an infection requiring systemic anti-infective therapy, open wounds, or has developed frequent acute or chronic infections during the past 12 weeks.
* Prior active tuberculosis.
* Total white blood cell count < 3.5 x 109/L at screening
* Neutrophil count of < 2.5 x 109/L at screening
* Platelet count of < 125 x 109/L at screening
* Hemoglobin < 8.0 g/dL at screening
* Abnormal liver function tests (AST/ALT > 1.5 x the upper limits of normal) at screening
* Abnormal renal function (serum creatinine > 1.5 x the upper limits of normal) at screening
* Prior treatment with any protein-based TNF inhibitor (e.g. etanercept, infliximab, PEG sTNF-RI, D2E7)
* Prior treatment with anakinra
* Receiving or has received any investigational drug within the previous 16 weeks or within at least 5 half-lives of any investigational drug, whichever is greater (or is currently using an investigational device)
* Received any intra-articular injections (e.g.. corticosteroids, hyaluronate preparations) or systemic corticosteroid injections within 4 weeks before the screening visit
* Requires analgesia other than paracetamol, NSAIDs, codeine, oxycodone, propoxyphene, tramadol, hydrocodone, or the combinations of these products (or equivalents)
* Subject (men or women of childbearing potential) is not using adequate contraceptive precautions as determined by the principal investigator
* Known allergy to E coli-derived products
* Not available for follow-up assessments
* Concerns for the subject's compliance with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2001-08; Primary Completion 2003-03 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Primary efficacy endpoint is the change from baseline at weeks 4, 26 and 52 in levels of select markers of inflammation (CD3 and CD 68) and destruction (MMP-1 and TIMP-1) in the synovium | up to 52 weeks
Primary safety endpoint is the crude and exposure adjusted subject incidence and nature, frequency, severity, relationship to treatment, and outcome of all adverse events | up to 52 weeks

SECONDARY OUTCOMES:
Secondary efficacy endpoints are change from baseline at week 4 and 52 in selected markers of bone and cartilage degradation and inflammation | up to 52 weeks
Secondary safety endpoints are changes from baseline in laboratory parameters | up to 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_25_IL-1RA_20000211.pdf
- See also: FDA-approved Drug Labeling — http://www.kineretrx.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com